CLINICAL TRIAL: NCT03766087
Title: Evaluation of the Benefits of Decompressive Craniectomy for Severe Traumatic Brain Injury in Children With Refractory Intracranial Hypertension
Brief Title: Decompressive Craniectomy for Severe Traumatic Brain Injury in Children With Refractory Intracranial Hypertension
Acronym: RANDECPED
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The authorization of the ethics committee lapses. No patients could be included in the study until the expiry of the ethics committee's authorization. The study never started
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-HPNCL-01
Record Dates: First submitted 2018-11-19; First posted 2018-12-06 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Hypertension Intracranial
MeSH Terms: conditions — Intracranial Hypertension | interventions — Decompressive Craniectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery group (Experimental): Decompressive craniectomy associated with optimal medical management of intracranial pressure.
  Interventions: Procedure: decompressive craniectomy
- conservative group (No Intervention): Optimal medical management of intracranial pressure only.

INTERVENTIONS:
Procedure: decompressive craniectomy — decompressive craniectomy is decompression at the supratentorial level that is achieved by removing part of the skull and by making an opening, in the dura mater (with or without plastic surgery), without compromising the venous sinus.
  Arms: surgery group

SUMMARY:
Severe traumatic brain injury (TBI) is the leading cause of mortality and severe disability in the pediatric population. The prognosis of these patients depends on the severity of the initial lesions but also on the effectiveness of the therapies used to prevent or at least limit secondary lesions mainly intracranial hypertension (HTIC).

The medical therapeutic strategy for the control of HTIC in children with TBI is well codified: starting with hyperosmolar therapy, then hyperventilation and ultimately the use of barbiturates to deepen sedation. However, these therapies are not devoid of adverse effects (hypernatremia, cerebral hypoxemia, systemic vasodilation) and, for some, their efficacy is diminished over time. When these treatments are insufficient to lower intracranial pressure (ICP), decompressive craniectomy is proposed. Decompressive craniectomy is used in a well-coded manner in malignant ischemic stroke in adults.

In TBI, to date, there are two randomized studies in adults and one in children but with a small number of patients, evaluating the benefit of decompressive craniectomy. None of them showed significantly superiority of the surgery compared to the maximal medication treatment on the functional prognosis in the medium term.

However, these studies have many biases, including a significant cross-over from the conservative treatment group to the surgery arm.

Nevertheless, the pediatric literature on the subject seems to yield better results on neurological prognosis in the long term. There are guidelines on the medical management of childhood TBI published by the National Institute of Health in 2012, which emphasize the need for controlled and randomized studies to define the place of decompressive craniectomy in children. That is why the investigators are proposing this national multicentre study.

DETAILED DESCRIPTION:
Severe Traumatic Brain Injury (STBI) constitutes the foremost cause of death and severe disability in the pediatric population. The severity of cranial trauma is evaluated by the Glasgow score. STBI corresponds with an initial Glasgow score of ≤ 8. The prognosis for patients with cranial trauma depends on the severity of the initial lesions, as well as the efficacy of the therapies applied to prevent, or at least limit, secondary lesions that are linked primarily to intracranial hypertension (ICH). Therapeutic treatments are based on the guidelines set by the Brain Trauma Foundation. These treatments mainly comprise heavy sedation known as "neurosedation" (maintaining hemodynamics, normothermia, hyperventilation, hyperosmolar therapy, and the administration of barbiturates).

When these therapies are not sufficiently effective, refractory ICH occurs, which is defined by a maximal value of intracranial pressure (ICP) as well as a minimal value for the Cerebral Perfusion Pressure (CPP), which corresponds to the Arterial Pressure (AP) minus the ICP (CPP=AP-ICP). Decompressive craniectomy (DC) may be used to treat refractory ICH. DC consists of removing part of the skull, which increase the "intracranial volume", thereby resulting in a decrease the ICP.

This surgical technique has been used systematically for several years to treat malignant ischemic stroke in adults. There have been three randomized studies to date of its use with STBI , of which only one was in regard to children. While decompressive craniectomy appears to decrease the ICP, no significant difference has been seen in adults in terms of the neurological outcomes when comparing patients who had an optimal medical management versus those who had this same treatment in conjunction with a decompressive craniectomy. Outcomes in children appear to be different, however, although the only randomized pediatric study had just 27 patients and the surgical technique that was used did not meet current standards. The other pediatric publications to date mostly involved series with limited numbers of cases and that hence do not allow conclusions to be drawn regarding the efficacy of craniectomy.

The latest guidelines underscore the need for controlled and randomized studies to establish the merits of decompressive craniectomy in children. This is why the investigators are proposing to undertake this study.

The main objective of this study is to compare decompressive craniectomy in association with an optimal medical management in children with Severe traumatic brain injury involving refractory intracranial hypertension, versus an optimal medical management only, in terms of the long-term (i.e. two year) functional neurological prognosis.

One of the secondary objectives is to compare the efficacy of decompressive craniectomy associated with an optimal medical management, versus an optimal medical management only, on the progression of the ICP in the 24 hours following randomization. The other secondary objectives will be to identify possible predictive factors of success two years after the decompressive craniectomy that are linked with characteristics of the patient, the type of trauma, the initial clinical condition, brain monitoring, radiological lesions, or surgical procedures.

For the main evaluation criterion, the investigators will use the functional neurological status of the patients at two years, which will be evaluated by the Glasgow Outcomes Scale-Extended Pediatric version (GOS E Peds). A satisfactory functional neurological status (i.e. success of the treatment) will be defined as a GOS E Peds ≥ 3.

The duration of the expected inclusions is two years, with a total duration for the study of four years and six months. In a prior retrospective study with 150 patients, the investigators found that the rate of favorable neurological progression at two years was approximately 60% of the patients after a decompressive craniectomy (publication in progress). Extrapolation of the main series in the literature allowed us to hypothesize that the favorable neurological progression rate at two years for patients in the control group was approximately 20%.

Thus, with a difference of 40% between the groups, a power of 80%, and an α risk=0.05; the number of patients required is 27 in each group. Based on our experience, in light of the very serious context of the pathology exhibited by these children and the risk of major sequelae, the investigators anticipate that few will be lost to follow-up.

The investigators estimate that approximately 90 children corresponding with the selection criteria are treated annually in the centers participating in the study. Based on our experience from prior studies in pediatric neurosurgery, the investigators assume the participation rate will be about 40%. It is hence reasonable to predict that inclusion over two years will yield 30 patients in each group.

Following admission to the resuscitation unit after a severe CT, all of the patients will undergo monitoring of their ICP and the patients will receive an initial treatment according to the relevant guidelines. If a patient lapses into a state of refractory ICH, compliance with the selection criteria will be checked, after which the study is explained to the parents by the anesthetist and the surgeon. If the patients agree to participate in the study, the patient is included in the study upon receipt of the signed informed consent, and the patients are randomized (by a centralized electronic randomization) into either the surgical group or the conservative group. The surgery will need to be performed in the 4 to 6 hours following the randomization. In both cases, the optimal medical management is also pursued.

Follow-up will initially be in the resuscitation unit and then in a hospital ward for the two groups. Visits at 1, 3, 6, 12, and 24 months will be scheduled along with recordings of the various clinical and radiological parameters, particularly with GOS E Peds scores at 12 and 24 months (the main criterion).

ELIGIBILITY:
Inclusion Criteria:

* Less than 18 years of age
* Severe traumatic brain injury (initial Glasgow coma scale < 9)
* Accidental trauma
* Refractory intracranial hypertension: ICP > 20 mmHg over 30 minutes for children more than one year of age and ICP > 15 mmHg over 30 minutes for children of less than one year of age.
* The patient must receive optimal medical management
* Affiliation with a social security scheme
* Signed informed consent is to be provided by the two holders of parental authority

Exclusion Criteria:

* Inflicted cranial trauma (e.g. shaken baby syndrome)
* Patients having an initial surgery for removal of an intracranial hemorrhagic collection of blood (e.g. a subdural hematoma, extradural hematoma, and intraparenchymal hematoma) for which the flap was not replaced.
* Pregnant patient

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
functional neurological status of the patients at 2 years | two years after surgery
  Functional neurological status (equating with success of the treatment) will be measure by the Glasgow Outcomes Scale-Extended Pediatric version.
  Extended GOS (GOSE) provides detailed categorization into eight categories by subdividing the categories of severe disability, moderate disability and good recovery into a lower and upper category. the GOSE range from 1 to 8 (Upper Good Recovery to Death).
  A score from 3 defines satisfactory functional neurological status. This threshold is selected as it equates to a moderate level of disability, that is to say a child that is autonomous in regard to daily activities and that is able to attend school

SECONDARY OUTCOMES:
Progression of the IntraCranial Pressure at 24 hours | 24 hours after inclusion
  the difference between the value of the ICP at 24 hours after inclusion and the value of the ICP at inclusion time
functional neurological status of the patients at 1 years | 1 year after inclusion
  Functional neurological status (equating with success of the treatment) will be measure by the Glasgow Outcomes Scale-Extended Pediatric version.
  A score from 3 defines satisfactory functional neurological status.
  SCORES:
  8 - Death 7 - Vegetative State 6 - Lower Severe Disability 5 - Upper Severe Disability 4 - Lower Moderate Disability 3 - Upper Moderate Disability 2 - Lower Good Recovery
  1 - Upper Good Recovery
Evaluation of the overall cognitive functioning | at 1 year and 2 years after inclusion
  neuropsychological assessment at one year and at two years using the Wechsler intelligence scales. the Wechsler intelligence scales are a Intelligence Quotient tests.
  Five standard tests are done to evaluate: the verbal comprehension index, the fluid reasoning index, the working memory index, and the processing speed index, as well as a total Intelligence Quotient.
  Classification of performance for scaled index scores are as follows:
  Below Average - scaled score 1 to 5 Low Average - scaled score 6 to 7 Average - scaled score 8 to 11 High Average - scaled score 12 to 13 Superior - 14 to 15 Very Superior - 16 to 20
  Descriptors of performance for standard WISC score ranges are as follows:
  Below Average - standard score below 79 Low Average - standard score 80 to 89 Average - 90 to 109 High Average - 110 to 119 Superior - 120 to 129 Very Superior - above 130
description of surgical parameters patients with successful craniectomy | at 2 years after craniectomy
  Collection of surgical parameters of the patient with successful surgery upon admission to resuscitation.
  The objective is to describe the predictive factors of successful craniectomy.
description of clinical parameters patients with successful craniectomy | at 2 years after craniectomy
  Collection of clinical parameters of the patient with successful surgery upon admission to resuscitation.
  The objective is to describe the predictive factors of successful craniectomy.
description of radiological parameters patients with successful craniectomy | at 2 years after craniectomy
  Collection of radiological parameters of the patient with successful surgery upon admission to resuscitation.
  The objective is to describe the predictive factors of successful craniectomy.
number of adverse events linked to surgery | from inclusion time to the end of patient participation, for about 2 years
  collection of adverse events linked to decompressive craniectomy and cranioplasty (infectious, hemorrhagic,cerebrospinal fluid )
Overall survival | at 3 months and 2 years post cranial trauma
  The survival time will be defined as the time between the date of the Crania Trauma and when death occurs from all causes combined.
Evaluation of quality of life | at 3 months, 1 years and 2 years
  measure of quality of life by Lansky scale, is a observational scoring system, in a range of 0-100. 0 represents unresponsive, and 100 represents full active, normal.

CONTACTS AND LOCATIONS:
Overall Officials: Michel LONJON, Pr, Principal Investigator — Hôpitaux Pédiatriques de Nice CHU-LENVAL
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No